CLINICAL TRIAL: NCT04518735
Title: Evolution of COVID-19 in Anticoagulated or Antiaggregated Patients
Brief Title: Evolution of COVID-19 in Anticoagulated or Antiaggregated Patients (CORONA Study)
Acronym: CORONA
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-24
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: Covid19; Oral anticoagulant; VKA; DOAC; Antiplatelet therapy; Heparin; Low molecular-weight heparin
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients on previous oral anticoagulant treatment: Patients receiving chronic anticoagulation with vitamin K antagonists (VKA, warfarin or acenocumarol) or with DOACs (dabigatran, rivaroxaban, apixaban or edoxaban) for any indication
  Interventions: Other: Antithrombotic Therapy (anticoagulant and/or antiplatelet) before admission for Covid19
- Patients on previous antiplatelet therapy: Patients receiving chronic antiplatelet therapy (aspirin, clopidogrel, prasugrel, ticagrelor, cangrelor, dipyridamol) for any indication
  Interventions: Other: Antithrombotic Therapy (anticoagulant and/or antiplatelet) before admission for Covid19
- Patients without antithrombotic therapy: Patients receiving nor chronic oral anticoagulation neither chronic antiplatelet therapy
  Interventions: Other: Antithrombotic Therapy (anticoagulant and/or antiplatelet) before admission for Covid19

INTERVENTIONS:
Other: Antithrombotic Therapy (anticoagulant and/or antiplatelet) before admission for Covid19 — Review of medical records during hospitalization and until day 28 post-entry to compare the clinical outcomes depending on previous antithrombotic therapy

SUMMARY:
CORONA is a retrospective, observational, one center study to investigate the clinical evolution (in terms of survival and thromboembolic complications) of patients on chronic treatment with anticoagulants or antiplatelet agents who are admitted to the hospital for COVID-19 compared with patients who do not receive anticoagulants or antiplatelet agents.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for COVID-19 at the Hospital de la Santa Creu i Sant Pau,
* Positive COVID-19 polymerase chain reaction test
* Length of stay more than 24 hours

Exclusion Criteria:

* No objective diagnose for COVID-19
* Outpatient
* Lenght of stay less than 24hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age and sex, suffering from Covid19 needing hospital admission more than 1 day for treatment and/or supportive care
Sampling Method: Non-Probability Sample
Enrollment: 1707 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality | From hospital admission to day 28
Transfer to the Intensive Care Unit (ICU) | From hospital admission to day 28

SECONDARY OUTCOMES:
Thromboembolic complications | From hospital admission to day 28
  Venous thromboembolism, ischemic stroke, myocardial infarction or periferal arterial thrombosis during hospitalization for Covid19
Major bleeding complications | From hospital admission to day 28
  Any bleeding complication grade 3 or 5 according BARC classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No